CLINICAL TRIAL: NCT00922454
Title: Acute Technical Outcomes of the Talent AAA Stent -Graft vs. Cook Zenith Stent- Graft: A Case-Control Study
Brief Title: Acute Technical Outcomes of the Talent Abdominal Aortic Aneurysm (AAA) Stent-Graft Versus Cook Zenith Stent-Graft
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Center for Vascular Awareness, Albany, New York (Other)
Responsible Party: Manish Mehta, MD, The Vascular Group, PLLC
Model: Crossover | Masking: None
Other Study IDs: 001
Record Dates: First submitted 2009-06-16; First posted 2009-06-17 (Estimated); Last update posted 2009-06-17 (Estimated); Status verified 2009-06

CONDITIONS: Abdominal Aortic Aneurysm
Keywords: patients will be matched based on AAA neck length and neck and iliac angulation
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Talent Stent-Graft (Experimental)
  Interventions: Procedure: Endovascular Repair of the abdominal aorta; Device: Talent Stent-Graft
- Cook Zenith Stent-Graft (Experimental)
  Interventions: Procedure: Endovascular Repair of the abdominal aorta; Device: Cook Zenith Stent-Graft

INTERVENTIONS:
Procedure: Endovascular Repair of the abdominal aorta — Patients will undergo or have undergone endovascular aneurysm repair which is minimally invasive approach using endoluminal placement of a stent graft.
  EVAR, CTA imaging, 1, 6 12 months post treatment.
Device: Cook Zenith Stent-Graft — Cook Zenith AAA Endovascular Graft
  Arms: Cook Zenith Stent-Graft
Device: Talent Stent-Graft — Talent AAA Abdominal Stent Graft System
  Arms: Talent Stent-Graft

SUMMARY:
The purpose of this study is to compare acute technical outcomes of the Talent AAA Stent Graft system versus Cook Zenith Endograft at two high volume institutions, Albany Medical Center and St. Peter's Hospital in Albany, NY.

The investigators are comparing the two devices as part of the evolution of endovascular repair (EVAR) for AAAs. The Zenith AAA Endovascular Graft received FDA approval on May 23, 2003, the Talent Abdominal Stent Graft System on April 15, 2008.

ELIGIBILITY:
Inclusion Criteria:

* subject with abdominal aortic aneurysm, with or without iliac involvement
* iliac/femoral access vessel morphology that is compatible with vascular access techniques, devices, and/or accessories

Exclusion Criteria:

* less than 18 years of age
* pregnant or lactating
* have contraindications for use of contrast medium or anticoagulation drugs
* are patients who have a condition that threatens to infect the graft
* are patients with sensitivities or allergies to the device materials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2009-06; Primary Completion 2011-06 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Acute technical success, successful exclusion of the aneurysm | one year

CONTACTS AND LOCATIONS:
Overall Officials: Manish Mehta, MD, MPH, Principal Investigator — The Vascular Group, PLLC
Locations (1):
- Albany Medical Center, 47 New Scotland Ave., Albany, New York, United States